CLINICAL TRIAL: NCT02755220
Title: A Prospective, Mutli-center, Open Lable, Single Arm Study to Evaluate the Safety and Effectiveness of Cingularbio® Heart Valve in Aortic/Mitral Valve Replacement Patients
Brief Title: Cingularbio® Heart Valve Clincial Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Cingularbio Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZBM-2015-01
Record Dates: First submitted 2016-04-24; First posted 2016-04-28 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2020-04

CONDITIONS: Diseases of Mitral and Aortic Valves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cingularbio® Heart valve (Experimental): the patients will replaced by artificial heart valve
  Interventions: Device: Cingularbio® Aortic valve replacement

INTERVENTIONS:
Device: Cingularbio® Aortic valve replacement — the patients will be replaced by Cingularbio heart valve

SUMMARY:
This study aimed to evaluate the safety and effectiveness of Cingularbio® heart valve in Aortic Valve Replacement and Mitral Valve Replacement in Chinese population

DETAILED DESCRIPTION:
single arm, 12 month follow up, mutile center, to assess the safety and effectiveness of Cingularbio® heart valve in Aortic Valve Replacement and Mitral Valve Replacement patients

ELIGIBILITY:
The inclusion criteria were as follows: 1) patient who had heart valve disease requiring a surgical replacement as indicated in the preoperative evaluation; 2) patient aged between 60-85 years; 3) patient whose preoperative heart function less than NYHA functional class IV; 4) patient who signed the informed consent before surgery; 5) patient who agrees to finish the follow-up. The exclusion criteria were as follows: 1) patient with prior valve replacement; 2) patient who requires concomitant tricuspid or pulmonary valve replacement; 3) patient who requires concomitant coronary artery bypass graft surgery; 4) patient with active infective endocarditis or drug abuse; 5) patient whose life time expectancy less than 12 months; 6) patient who was unable to follow anticoagulation treatment.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
device related adverse valve events | 12 month
  device related events including Thromboembolism, Valve thrombosis,Major hemorrhage, Major paravalvular leak

SECONDARY OUTCOMES:
rate of procedural success | post-operative
  device implant success
the difference between baseline and 1 year in Effective orifice area (EOA) | 1year
  the difference between baseline and 1 year in Effective orifice area (EOA) in echocardiographic hemodynamic
the difference between baseline and 1 year in pressure gradient (PG) | 1year
  the difference between baseline and 1 year in pressure gradient (PG) in echocardiographic hemodynamic
the difference between baseline and 1 year in Peak aortic valve velocity | 1year
  the difference between baseline and 1 year in Peak aortic valve velocity in echocardiographic hemodynamic
improvement in NYHA functional class | 1year
  the NYHA score between baseline and 1 year
mortality | 1 year
  the mortality rate at 1 year
structural valve deterioration | 1 year
  the SVD rate at 1 year
reoperation | 1 year
  the reoperation rate at 1 year
valve-related adverse events | 1 year
  all valve related AEs (not primary endpoint events) at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: chunsheng wang, Principal Investigator — Fudan University
Locations (5):
- Cardiale Heelkunde, Leuven, Belgium
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China
- Poland (3):
  - Klinika Kardiochirurgii, Katowice
  - Klinika Kardiochirurgii, Krakow
  - Klinika Kardiochirurgii, Warsaw

IPD SHARING:
Plan to Share IPD: No
the publication will be started after study close out